CLINICAL TRIAL: NCT01916993
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Single Dose of NBI-98854 in Subjects With Mild, Moderate, or Severe Hepatic Insufficiency
Brief Title: Safety, Tolerability, and Pharmacokinetics of a Single Dose of NBI-98854 in Subjects With Mild,Moderate, or Severe Hepatic Insufficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NBI-98854-1303
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Safety, Tolerability, and PK of NBI-98854 in Hepatically Impaired Subjects
MeSH Terms: interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy Volunteers (Experimental): single dose of NBI-98854 50 mg capsule
  Interventions: Drug: NBI-98854 50 mg capsule
- Mild Hepatic Impairment (Experimental): single dose of NBI-98854 50 mg capsule
  Interventions: Drug: NBI-98854 50 mg capsule
- Moderate Hepatic Impairment (Experimental): single dose of NBI-98854 50 mg capsule
  Interventions: Drug: NBI-98854 50 mg capsule
- Severe Hepatic Impairment (Experimental): single dose of NBI-98854 50 mg capsule
  Interventions: Drug: NBI-98854 50 mg capsule

INTERVENTIONS:
Drug: NBI-98854 50 mg capsule

SUMMARY:
The purpose of this research study is to: test the safety, tolerability, and pharmacokinetics (PK testing, the study of how the body absorbs, distributes, breaks down and eliminates a drug) of a single dose of the investigational study drug NBI-98854 in subjects with normal hepatic function or mild, moderate, or severe hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age.
* Healthy volunteers must be in good general health.
* Subjects with hepatic impairment must be judged to be in stable condition.
* Subjects of childbearing potential must agree to use hormonal or two forms of nonhormonal birth control during the study.
* Female subjects must not be pregnant, given birth within 1 year of study start, or breastfeeding.
* Have a body mass index (BMI) of 18 to 40 kg/m2 (both inclusive).

Exclusion Criteria:

* Report more than two alcoholic beverages daily or more than 14 alcoholic beverages weekly withing 7 days of study start.
* Have a known history of neuroleptic malignant syndrome.
* Have a positive human immunodeficiency virus (HIV) antibody result at screening or have a history of positive result.
* Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study.
* Have an allergy, hypersensitivity, or intolerance to tetrabenazine.
* Had a blood loss greater than or equal to 500 mL or donated blood within 56 days of study start.
* Have had previous exposure with NBI-98854.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of plasma concentrations of NBI-98854 and metabolites following administration of NBI-98854 | 45 minutes prior to NBI-98854 dosing, and 15, 30, 45 minutes, and 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, and 120 hours postdose
Number of Participants with Adverse Events following dosing with NBI-98854 | Up to 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD, Study Director — Neurocrine Biosciences
Locations (3):
- United States (3):
  - DaVita Clinical Research, Lakewood, Colorado
  - Orlando Clinical Research Center, Orlando, Florida
  - Davita Clinical Research, Minneapolis, Minnesota